CLINICAL TRIAL: NCT00096850
Title: Safety, Tolerability, and Pharmacokinetic Interactions of Atazanavir and Rifampin in Healthy Volunteers
Brief Title: Safety, Tolerability, and Blood Levels of Ritonavir-Boosted Atazanavir and Rifampin When Taken Together in HIV Uninfected Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5213; 10021 (Registry Identifier: DAIDS ES); ACTG A5213
Record Dates: First submitted 2004-11-16; First posted 2004-11-17 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV Seronegativity; Antitubercular agents
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Atazanavir Sulfate; Rifampin; Ritonavir

ARMS (1):
- 1 (Experimental): From Days 1 to 8, participants will receive 600 mg RIF every 24 hours. From Days 9 to 19, participants will receive 300 mg ATV and 100 mg RTV every 12 hours and 600 mg RIF every 24 hours. From Days 20 to 27, participants will receive 400 mg ATV and 100 mg RTV every 12 hours and 600 mg RIF every 24 hours.
  Interventions: Drug: Atazanavir; Drug: Rifampin; Drug: Ritonavir

INTERVENTIONS:
Drug: Atazanavir — From Days 9 to 19, participants will receive a 300 mg tablet orally daily. From Days 20 to 27, participants will receive a 400 mg tablet orally daily.
  Other Names: ATV
Drug: Rifampin — From Days 1 to 27, participants will receive a 600 mg tablet orally daily.
  Other Names: RIF
Drug: Ritonavir — From Days 9 to 19, participants will receive a 100 mg tablet orally daily. From Days 20 to 27, participants will receive a 100 mg tablet orally twice daily.
  Other Names: RTV

SUMMARY:
Rifampin (RIF) is used for the treatment of tuberculosis (TB), an infectious disease that affects many people with HIV. RIF was shown to lower concentrations and decrease the effectiveness of some anti-HIV drugs, including the HIV protease inhibitor (PI) atazanavir (ATV) boosted with ritonavir (RTV). The purpose of this study is to determine the interactions between RTV-boosted ATV and evaluate the safety and tolerability of giving these drugs together in HIV uninfected adults.

DETAILED DESCRIPTION:
TB is common in resource-limited countries, and people infected with HIV are especially at risk for TB infection. The antituberculous drug RIF lowers plasma concentrations of PIs by increasing the activity of enzymes responsible for PI breakdown. RIF has been shown to reduce PI effectiveness, a particular concern for HIV infected patients who are also being treated for TB. RTV has been shown to delay the plasma clearance of ATV and increase the plasma half-life of ATV. This study will evaluate the safety, tolerability, and pharmacokinetic (PK) interactions of RTV-boosted ATV, taken concurrently with RIF in HIV uninfected people.

Medical and medication history, a complete physical exam, blood collection, and an electrocardiogram (ECG) will occur at screening. Participants will be enrolled in this study for 41 to 58 days; there will be 3 dosing periods. From Days 1 to 8, participants will receive 600 mg RIF every 24 hours. From Days 9 to 19, participants will receive 300 mg ATV and 100 mg RTV every 12 hours and 600 mg RIF every 24 hours. From Days 20 to 27, participants will receive 400 mg ATV and 100 mg RTV every 12 hours and 600 mg RIF every 24 hours. Study visits will occur at entry; at Days 5, 8, 11, 14, 19, 23, and 27; and at an additional visit between Days 41 and 48. Blood and urine collection will occur at all visits. A targeted physical exam, an ECG, and blood collection for PK analysis will occur at Days 8, 19, and 27.

ELIGIBILITY:
Note: As of 11/27/06, enrollment into Version 1.0 of the study is now closed. Any new study participants will enroll under Version 2.0.

Inclusion Criteria:

* HIV uninfected
* Normal creatinine clearance
* Willing to use acceptable means of contraception during the study and for at least 6 weeks after stopping study medications

Exclusion Criteria:

* Using or anticipating use of certain medications, including any medication metabolized by CYP3A
* Active drug use or dependence that, in the opinion of the investigator, may interfere with the study
* Cannot stop consuming alcoholic beverages, grapefruit, or grapefruit juice for the duration of the study
* Cannot stop consuming coffee or caffeine-containing products for 12 hours prior to Day 8, 19, and 27 PK studies
* Serious illness that, in the opinion of the investigator, may interfere with the study
* Hospitalization for any reason within 14 days prior to study entry
* History of hypersensitivity to study drugs or their formulations
* Active or previous history of cardiovascular, kidney, liver, blood, neurologic, gastrointestinal, psychiatric, endocrine, or immunologic disease. Patients with chronic illnesses such as hypertension, coronary heart disease, arthritis, diabetes, or chronic gastrointestinal conditions that may affect drug absorption are also excluded.
* ECG showing first-degree or greater heart block or a QT interval greater than 440 msec within 30 days of study entry
* Previous participation in this study
* Pregnancy or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of ritonavir (RTV)-boosted ATV when administered concurrently with RIF | Throughout study
Safety and tolerability of RTV-boosted ATV when coadministered with RIF | Throughout study

SECONDARY OUTCOMES:
Pharmacokinetics of RIF | Throughout study
Copy number of cellular drug transporter RNA in peripheral blood mononuclear cells (PBMCs) | Throughout study
UDP-glucuronosyltransferase (UGT)-1A1 genotype | At study entry
Serum bilirubin concentration | Throughout study
urine thromboxane and prostacyclin concentrations | At study entry and first PK visit

CONTACTS AND LOCATIONS:
Overall Officials: David W. Haas, MD, Study Chair — Infectious Diseases, Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Stanford CRS, Palo Alto, California
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee

REFERENCES:
- [Background] Finch CK, Chrisman CR, Baciewicz AM, Self TH. Rifampin and rifabutin drug interactions: an update. Arch Intern Med. 2002 May 13;162(9):985-92. doi: 10.1001/archinte.162.9.985. PMID 11996607
- [Background] Fujiwara PI, Clevenbergh P, Dlodlo RA. Management of adults living with HIV/AIDS in low-income, high-burden settings, with special reference to persons with tuberculosis. Int J Tuberc Lung Dis. 2005 Sep;9(9):946-58. PMID 16158886
- [Background] Kashuba AD. Drug-drug interactions and the pharmacotherapy of HIV infection. Top HIV Med. 2005 Jun-Jul;13(2):64-9. PMID 16082056
- [Background] Musial BL, Chojnacki JK, Coleman CI. Atazanavir: a new protease inhibitor to treat HIV infection. Am J Health Syst Pharm. 2004 Jul 1;61(13):1365-74. doi: 10.1093/ajhp/61.13.1365. PMID 15287232
- [Background] Orrick JJ, Steinhart CR. Atazanavir. Ann Pharmacother. 2004 Oct;38(10):1664-74. doi: 10.1345/aph.1D394. Epub 2004 Sep 7. PMID 15353575
- [Result] Acosta EP, Kendall MA, Gerber JG, Alston-Smith B, Koletar SL, Zolopa AR, Agarwala S, Child M, Bertz R, Hosey L, Haas DW. Effect of concomitantly administered rifampin on the pharmacokinetics and safety of atazanavir administered twice daily. Antimicrob Agents Chemother. 2007 Sep;51(9):3104-10. doi: 10.1128/AAC.00341-07. Epub 2007 Jun 18. PMID 17576825